CLINICAL TRIAL: NCT02222922
Title: A FIRST-IN-HUMAN PHASE 1, DOSE ESCALATION, SAFETY AND PHARMACOKINETIC STUDY OF PF-06647020 IN ADULT PATIENTS WITH ADVANCED SOLID TUMORS
Brief Title: A Study Of PF-06647020 For Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: B7661001; 2014-003296-36 (EudraCT Number)
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Neoplasms
Keywords: ADC; PF-06647020; solid tumors; tumors; neoplasm metastasis; TNBC; triple negative breast cancer; NSCLC; non small cell lung cancer; advanced metastatic breast cancer; ovarian cancer; OVCA
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms | interventions — Fluconazole; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PF-06647020 Q3W (Experimental): Investigational drug infused over 60 minutes once every 21 days.
  Interventions: Drug: PF-06647020 Q3W
- Drug-drug interaction (DDI) (Experimental): PF-06647020 combined with fluconazole
  Interventions: Drug: fluconazole
- PF-06647020 Q2W (Experimental): Investigational drug infused over 60 minutes once every 14 days (28 day cycle)
  Interventions: Drug: PF-06647020 Q2W
- PF-06647020 combined with Avelumab (Experimental): PF-06647020 combined with Avelumab administered by infusion
  Interventions: Drug: PF-06647020 combined with Avelumab

INTERVENTIONS:
Drug: PF-06647020 Q3W — Part 1: PF-06647020 will be administered intravenously every 21 days in cohorts of 2-4 patients starting at a dose of 0.20mg/kg. Increases in dose will continue until MTD is determined.
  Part 2: Patients with triple negative breast cancer (pre-selected for PTK7 moderately high to high expression), non small cell lung cancer (pre-selected with moderate to high PTK7 expression) and ovarian cancer patients (unselected for PTK7 expression) will be treated at the MTD or Recommended Phase 2 Dose selected in Part 1.
  Arms: PF-06647020 Q3W
Drug: fluconazole — combination drug used for drug-drug interaction sub-study
  Arms: Drug-drug interaction (DDI)
Drug: PF-06647020 Q2W — Part 1: PF-06647020 will be administered intravenously every 14 days in cohorts of 2-4 patients starting at a dose of 2.1 mg/kg. Increases in dose will continue until MTD is determined.
  Part 2: Patients with non-small cell lung cancer (pre-selected for PTK7 moderate to high expression and ovarian cancer patients (unselected for PTK7 expression) will be treated at the MTD or Recommended Phase 2 Dose selected in Part 1.
  Arms: PF-06647020 Q2W
Drug: PF-06647020 combined with Avelumab — Part 2: Patients with ovarian cancer (unselected for PTK7 expression) will be treated with PF-0664702 plus Avelumab.
  Arms: PF-06647020 combined with Avelumab

SUMMARY:
To assess the safety and tolerability at increasing dose levels of PF-06647020 in patients with advanced solid tumors in order to determine the maximum tolerated dose and select the recommended Phase 2 dose.

ELIGIBILITY:
Q2W Inclusion Criteria:

* Diagnosis of platinum resistant or refractory OVCA having received 2 or fewer prior lines, or recurrent advanced NSCLC having received 3 or fewer prior lines
* Performance Status of 0, 1, or 2
* Adequate bone marrow, kidney, and liver function

Q2W Exclusion Criteria:

* OVCA pts excluded with any of the following: non-epithelial, including malignant mixed mullerian tumors, unresolved bowel obstruction
* Brain metastases requiring steroids
* Major surgery, radiation therapy, or systemic anti-cancer therapy within 4 weeks of study treatment start
* Active and clinically significant bacterial, fungal, or viral infection

Q3W Inclusion Criteria:

* Diagnosis of solid tumor that is advanced/metastatic and resistant to standard therapy or for whom no standard therapy is available
* Performance Status of 0 or 1
* Adequate bone marrow, kidney, and liver function
* Part 2 includes ovarian cancer, target expressing triple negative breast cancer and non small cell lung cancer patients

Q3W Exclusion Criteria:

* OVCA pts excluded with any of the following: non-epithelial, including malignant mixed mullerian tumors, prior radiotherapy to pelvis/abdomen, pts with CA-125 only disease, unresolved bowel obstruction
* Brain metastases requiring steroids
* Major surgery, radiation therapy, or systemic anti-cancer therapy within 4 weeks of study treatment start
* Active and clinically significant bacterial, fungal, or viral infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2014-10-17 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Scottsdale Healthcare Hospitals DBA HonorHealth, Scottsdale, Arizona
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Stanford Cancer Center, Stanford, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Chicago Medicine, Chicago, Illinois
  - START Midwest, Grand Rapids, Michigan
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - Inova Fairfax Hospital Woodburn GYN Infusion Center, Annandale, Virginia
  - Mid Atlantic Gynecologic Oncology and Pelvic Surgery Associates (MAGOPSA), Annandale, Virginia
  - Fairfax Radiological Consultants, Fairfax, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Loudon Hospital, Leesburg, Virginia
- Spain (2):
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Johnson M, El-Khoueiry A, Hafez N, Lakhani N, Mamdani H, Rodon J, Sanborn RE, Garcia-Corbacho J, Boni V, Stroh M, Hannah AL, Wang S, Castro H, Spira A. Phase I, First-in-Human Study of the Probody Therapeutic CX-2029 in Adults with Advanced Solid Tumor Malignancies. Clin Cancer Res. 2021 Aug 15;27(16):4521-4530. doi: 10.1158/1078-0432.CCR-21-0194. Epub 2021 Jun 3. PMID 34083236
- [Derived] Maitland ML, Sachdev JC, Sharma MR, Moreno V, Boni V, Kummar S, Stringer-Reasor E, Lakhani N, Moreau AR, Xuan D, Li R, Powell EL, Jackson-Fisher A, Bowers M, Alekar S, Xin X, Tolcher AW, Calvo E. First-in-Human Study of PF-06647020 (Cofetuzumab Pelidotin), an Antibody-Drug Conjugate Targeting Protein Tyrosine Kinase 7, in Advanced Solid Tumors. Clin Cancer Res. 2021 Aug 15;27(16):4511-4520. doi: 10.1158/1078-0432.CCR-20-3757. Epub 2021 Jun 3. PMID 34083232
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7661001&StudyName=A%20Study%20Of%20PF-06647020%20For%20Adult%20Patients%20With%20Advanced%20Solid%20Tumors%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Once every 3 weeks (Q3W) Regimen: A total of 113 participants were enrolled to study treatments and 1 participant in the PF-06647020 2.1 mg/kg treatment group didn't receive any study treatment.
  Once every 2 weeks (Q2W) Regimen: A total of 25 participants were enrolled to study treatments and all were treated with study drug.
Groups:
- PF-06647020 0.2 mg/kg (Q3W Regimen): Participants received PF-06647020 at 0.2 mg/kg on Day 1 of each 21-day cycle as an intravenous (IV) infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination. The maximum duration of treatment in this arm was approximately 4.8 months.
- PF-06647020 0.5 mg/kg (Q3W Regimen): Participants received PF-06647020 at 0.5 mg/kg on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination. The maximum duration of treatment in this arm was approximately 0.7 months.
- PF-06647020 1.25 mg/kg (Q3W Regimen): Participants received PF-06647020 at 1.25 mg/kg on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination. The maximum duration of treatment in this arm was approximately 3.5 months.
- PF-06647020 2.1 mg/kg (Q3W Regimen): Participants received PF-06647020 at 2.1 mg/kg on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination. The maximum duration of treatment in this arm was approximately 8.6 months.
- PF-06647020 2.8 mg/kg (Q3W Regimen): Participants received PF-06647020 at 2.8 mg/kg on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination. The maximum duration of treatment in this arm was approximately 30 months.
- PF-06647020 3.7 mg/kg (Q3W Regimen): Participants received PF-06647020 at 3.7 mg/kg on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination. The maximum duration of treatment in this arm was approximately 8.6 months.
- PF-06647020 2.1 mg/kg (Q2W Regimen): Participants received PF-06647020 at 2.1 mg/kg on Days 1 and 15 of each 28-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination. The maximum duration of treatment in this arm was approximately 3.2 months.
- PF-06647020 2.8 mg/kg (Q2W Regimen): Participants received PF-06647020 at 2.8 mg/kg on Days 1 and 15 of each 28-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination. The maximum duration of treatment in this arm was approximately 16.4 months.
- PF-06647020 3.2 mg/kg (Q2W Regimen): Participants received PF-06647020 at 3.2 mg/kg on Days 1 and 15 of each 28-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination. The maximum duration of treatment in this arm was approximately 17.1 months.
Period: Overall Study
Arm/Group | PF-06647020 0.2 mg/kg (Q3W Regimen) | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Started | 2 | 2 | 2 | 5 | 96 | 6 | 3 | 10 | 12
Received Treatment | 2 | 2 | 2 | 4 | 96 | 6 | 3 | 10 | 12
Completed | 1 | 2 | 1 | 2 | 58 | 3 | 1 | 6 | 6
Not Completed | 1 | 0 | 1 | 3 | 38 | 3 | 2 | 4 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 13 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 9 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 2 | 10 | 2 | 2 | 4 | 1
Not completed — Participant refused further follow-up | 1 | 0 | 0 | 1 | 6 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all enrolled participants who received at least 1 full or partial dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06647020 0.2 mg/kg (Q3W Regimen) | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen) | Total
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 6 | 3 | 10 | 12 | 137
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Since the Q3W and Q2W regimens were assessed independently for the purpose of this study, therefore, baseline data for these regimens are presented in separate rows.
  Years
    Q3W Regimen: number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 6 | 0 | 0 | 0 | 112
    Q3W Regimen | 73.0 (2.8) | 57.5 (14.8) | 61.0 (2.8) | 55.0 (13.6) | 58.1 (11.8) | 59.5 (8.4) |  |  |  | 58.4 (11.6)
    Q2W Regimen: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 10 | 12 | 25
    Q2W Regimen |  |  |  |  |  |  | 64.0 (2.6) | 65.5 (8.9) | 65.6 (8.0) | 65.4 (7.8)
Age, Customized [Count of Participants; unit: Participants] — Population: Since the Q3W and Q2W regimens were assessed independently for the purpose of this study, therefore, baseline data for these regimens are presented in separate rows.
  Participants
    < 18 (Q3W Regimen): number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 6 | 0 | 0 | 0 | 112
    < 18 (Q3W Regimen) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    18-44 (Q3W Regimen): number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 6 | 0 | 0 | 0 | 112
    18-44 (Q3W Regimen) | 0 | 0 | 0 | 0 | 16 | 0 | 0 | 0 | 0 | 16
    45-64 (Q3W Regimen): number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 6 | 0 | 0 | 0 | 112
    45-64 (Q3W Regimen) | 0 | 1 | 2 | 3 | 49 | 4 | 0 | 0 | 0 | 59
    >= 65 (Q3W Regimen): number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 6 | 0 | 0 | 0 | 112
    >= 65 (Q3W Regimen) | 2 | 1 | 0 | 1 | 31 | 2 | 0 | 0 | 0 | 37
    < 18 (Q2W Regimen): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 10 | 12 | 25
    < 18 (Q2W Regimen) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    18-44 (Q2W Regimen): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 10 | 12 | 25
    18-44 (Q2W Regimen) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    45-64 (Q2W Regimen): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 10 | 12 | 25
    45-64 (Q2W Regimen) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 6 | 12
    >= 65 (Q2W Regimen): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 10 | 12 | 25
    >= 65 (Q2W Regimen) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Since the Q3W and Q2W regimens were assessed independently for the purpose of this study, therefore, baseline data for these regimens are presented in separate rows.
  Participants
    Q3W Regimen: number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 6 | 0 | 0 | 0 | 112
    Q3W Regimen: Female | 2 | 1 | 1 | 3 | 80 | 5 | 0 | 0 | 0 | 92
    Q3W Regimen: Male | 0 | 1 | 1 | 1 | 16 | 1 | 0 | 0 | 0 | 20
    Q2W Regimen: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 10 | 12 | 25
    Q2W Regimen: Female | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 10 | 11 | 24
    Q2W Regimen: Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Since the Q3W and Q2W regimens were assessed independently for the purpose of this study, therefore, baseline data for these regimens are presented in separate rows.
  Participants
    Q3W Regimen: number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 6 | 0 | 0 | 0 | 112
    Q3W Regimen: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Q3W Regimen: Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Q3W Regimen: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Q3W Regimen: Black or African American | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 6
    Q3W Regimen: White | 2 | 2 | 2 | 3 | 88 | 6 | 0 | 0 | 0 | 103
    Q3W Regimen: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Q3W Regimen: Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
    Q2W Regimen: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 10 | 12 | 25
    Q2W Regimen: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Q2W Regimen: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Q2W Regimen: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Q2W Regimen: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Q2W Regimen: White | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 8 | 11 | 21
    Q2W Regimen: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Q2W Regimen: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Weight Continuous [Mean (Standard Deviation); unit: kilogram (kg)] — Population: Since the Q3W and Q2W regimens were assessed independently for the purpose of this study, therefore, baseline data for these regimens are presented in separate rows.
  kilogram (kg)
    Q3W Regimen: number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 6 | 0 | 0 | 0 | 112
    Q3W Regimen | 49.2 (10.2) | 68.8 (21.9) | 68.7 (5.2) | 80.7 (27.3) | 69.9 (16.4) | 72.2 (14.2) |  |  |  | 70.0 (16.6)
    Q2W Regimen: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 10 | 12 | 25
    Q2W Regimen |  |  |  |  |  |  | 68.4 (23.8) | 78.1 (25.5) | 68.3 (22.5) | 72.3 (23.4)
Body Mass Index (BMI) Continuous [Mean (Standard Deviation); unit: kg/m^2] — Population: Since the Q3W and Q2W regimens were assessed independently for the purpose of this study, therefore, baseline data for these regimens are presented in separate rows.
  kg/m^2
    Q3W Regimen: number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 6 | 0 | 0 | 0 | 112
    Q3W Regimen | 18.3 (2.0) | 22.7 (2.7) | 23.6 (2.0) | 27.6 (7.7) | 25.6 (5.5) | 26.2 (4.7) |  |  |  | 25.5 (5.5)
    Q2W Regimen: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 10 | 12 | 25
    Q2W Regimen |  |  |  |  |  |  | 24.9 (7.1) | 29.9 (9.1) | 25.6 (8.8) | 27.2 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) - Q3W Regimen
Description: A DLT was any of the following adverse events(AEs) in the first cycle of treatment (within 21 days of first dose or until participant received second infusion if there were treatment delays). (1)Hematologic: including Grade 4 neutropenia lasting >7 days; Febrile neutropenia; Grade >=3 neutropenic infection; Grade 4 anemia; Grade >=3 thrombocytopenia with clinically significant bleeding. (2) Hepatic, including Grade >=3 serum bilirubin, hepatic transaminase or alkaline phosphatase; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >=3.0 x upper limit of normal (ULN) concurrent with elevation in bilirubin >=2.0 x ULN; (3) Grade >=3 non-hematologic, non-hepatic major organ toxicities; delayed by >2 weeks in receiving the next scheduled cycle due to persisting toxicities attributable to PF-06647020. A participant was on study for at least 21 days to be evaluable for DLT observation, and could be replaced if they terminated study participation earlier than 21 days.
Time Frame: First Cycle, Day 1 up to Day 21
Population: Participants enrolled in the dose escalation phase in Q3W regimen who received at least 1 dose of study medication and who did not have major treatment deviations during first cycle with a baseline disease assessment and at least 1 post-baseline disease assessment.
Measure: Count of Participants; unit: Participants
Groups:
- PF-06647020 0.2 mg/kg（Q3W Regimen）: Participants enrolled in the dose escalation phase received PF-06647020 at 0.2 mg/kg on Day 1 of each 21-day cycle as an intravenous (IV) infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
- PF-06647020 0.5 mg/kg (Q3W Regimen): Participants enrolled in the dose escalation phase received PF-06647020 at 0.5 mg/kg on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
- PF-06647020 1.25 mg/kg (Q3W Regimen): Participants enrolled in the dose escalation phase received PF-06647020 at 1.25 mg/kg on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
- PF-06647020 2.1 mg/kg (Q3W Regimen): Participants enrolled in the dose escalation phase received PF-06647020 at 2.1 mg/kg on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
- PF-06647020 2.8 mg/kg (Q3W Regimen): Participants enrolled in the dose escalation phase received PF-06647020 at 2.8 mg/kg on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
- PF-06647020 3.7 mg/kg (Q3W Regimen): Participants enrolled in the dose escalation phase received PF-06647020 at 3.7 mg/kg on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 15 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 2

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) - Q3W Regimen (All-Causality)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study medication.
Time Frame: From the time the participant took the first dose of study medication through the participant's last visit. (approximately 32 months)
Population: All participants enrolled in Q3W regimen who received at least 1 full or partial dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- PF-06647020 0.2 mg/kg（Q3W Regimen）: Participants received PF-06647020 at 0.2 mg/kg on Day 1 of each 21-day cycle as an intravenous (IV) infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination. The maximum duration of treatment in this arm was approximately 4.8 months.
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 6
Participants
  AEs | 2 | 2 | 2 | 4 | 96 | 6
  SAEs | 0 | 0 | 0 | 1 | 33 | 2

3. Primary Outcome: Number of Participants With Treatment-Emergent AEs - Q3W Regimen (Treatment-Related)
Description: A treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study medication.
Time Frame: as for outcome 2
Population: All participants enrolled in Q3W regimen who received at least 1 full or partial dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 6
Participants
  AEs | 1 | 1 | 1 | 4 | 84 | 5
  SAEs | 0 | 0 | 0 | 1 | 9 | 0

4. Primary Outcome: Number of Participants With Treatment-Emergent AEs Categorized by Seriousness - Q3W Regimen (All-Causality and Treatment-Related)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study medication. All AEs were graded by the investigator according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Grade 1 AEs are mild AEs; Grade 2 AEs are moderate AEs; Grade 3 AEs are severe AEs, Grade 4 AEs are life-threatening consequences and Grade 5 AEs are deaths related to AEs. Each AE was counted once for the participant in the most severe severity.
Time Frame: as for outcome 2
Population: All participants enrolled in Q3W regimen who received at least 1 full or partial dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 6
Participants
  Grade 1 (all-causality) | 0 | 0 | 1 | 1 | 6 | 0
  Grade 2 (all-causality) | 1 | 2 | 0 | 2 | 18 | 1
  Grade 3 (all-causality) | 1 | 0 | 1 | 1 | 49 | 5
  Grade 4 (all-causality) | 0 | 0 | 0 | 0 | 14 | 0
  Grade 5 (all-causality) | 0 | 0 | 0 | 0 | 9 | 0
  Missing or Unknown (all-causality) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 1 (treatment-related) | 0 | 1 | 1 | 1 | 23 | 1
  Grade 2 (treatment-related) | 0 | 0 | 0 | 3 | 21 | 1
  Grade 3 (treatment-related) | 1 | 0 | 0 | 0 | 28 | 3
  Grade 4 (treatment-related) | 0 | 0 | 0 | 0 | 12 | 0
  Grade 5 (treatment-related) | 0 | 0 | 0 | 0 | 0 | 0
  Missing or Unknown (treatment-related) | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Hematology Laboratory Abnormalities (All Cycles) - Q3W Regimen
Description: Participants who experienced hematology laboratory test abnormalities were summarized according to worst toxicity grade observed for each hematology laboratory test. Laboratory abnormalities were graded by NCI CTCAE version 4.03. This outcome measure calculated the number of participants with hematology laboratory abnormalities that were shifted from <=Grade 2 at baseline to Grade 3 or above, including the following parameters: absolute neutrophils, lymphopenia, white blood cell, anemia, platelets.
Time Frame: From baseline to end of treatment (approximately 32 months).
Population: All participants enrolled in Q3W regimen who received at least 1 full or partial dose of study medication and had at least 1 observation of the given hematology laboratory test.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 5
Participants
  Absolute neutrophils | 0 | 0 | 0 | 1 | 28 | 2
  Lymphopenia | 1 | 1 | 0 | 0 | 21 | 2
  White blood cells | 0 | 0 | 0 | 0 | 18 | 1
  Anemia | 0 | 0 | 0 | 0 | 2 | 0
  Platelets | 0 | 0 | 0 | 0 | 2 | 0

6. Primary Outcome: Number of Participants With Chemistry Laboratory Abnormalities (All Cycles) - Q3W Regimen
Description: Participants who experienced chemistry laboratory test abnormalities were summarized according to worst toxicity grade observed for each chemistry laboratory test. Laboratory abnormalities were graded by NCI CTCAE version 4.03. This outcome measure calculated the number of participants with chemistry laboratory abnormalities that were shifted from <=Grade 2 at baseline to Grade 3 or above, including the following parameters: hypokalemia, hypophosphatemia, aspartate aminotransferase, hyperglycemia, alkaline phosphatase, hyponatremia, alanine aminotransferase, hypoalbuminemia, total bilirubin, hypercalcemia, hypomagnesemia , creatinine, gamma glutamyl transferase, hypocalcemia.
Time Frame: From baseline to end of treatment (approximately 32 months).
Population: All participants enrolled in Q3W who received at least 1 full or partial dose of study medication and had at least 1 observation of the given chemistry laboratory test.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 5
Participants
  Hypokalemia | 0 | 0 | 0 | 0 | 8 | 1
  Hypophosphatemia | 0 | 0 | 0 | 0 | 8 | 1
  Aspartate aminotransferase | 0 | 0 | 0 | 0 | 6 | 0
  Hyperglycemia | 0 | 0 | 0 | 0 | 6 | 0
  Alkaline phosphatase | 0 | 0 | 0 | 0 | 6 | 0
  Hyponatremia | 1 | 0 | 0 | 0 | 4 | 0
  Alanine aminotransferase | 0 | 0 | 0 | 0 | 4 | 0
  Hypoalbuminemia | 0 | 0 | 0 | 0 | 3 | 0
  Total bilirubin | 0 | 0 | 0 | 0 | 2 | 0
  Hypercalcemia | 0 | 0 | 0 | 0 | 2 | 0
  Hypomagnesemia | 0 | 0 | 0 | 0 | 2 | 0
  Creatinine | 0 | 0 | 0 | 0 | 1 | 0
  Gamma glutamyl transferase | 0 | 0 | 0 | 0 | 1 | 0
  Hypocalcemia | 0 | 0 | 0 | 0 | 1 | 0

7. Primary Outcome: Number of Participants With Urinalysis Laboratory Abnormalities (All Cycles) - Q3W Regimen
Description: Participants who experienced urinalysis laboratory test abnormalities were summarized according to worst toxicity grade observed for each urinalysis laboratory test. Laboratory abnormalities were graded by NCI CTCAE version 4.03. This outcome measure calculated the number of participants with urinalysis laboratory abnormalities that were shifted from <=Grade 2 at baseline to Grade 3 or above.
Time Frame: From baseline to end of treatment (approximately 32 months).
Population: All participants enrolled in Q3W regimen who received at least 1 full or partial dose of study medication and had at least 1 observation of the given urinalysis laboratory test.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 93 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Coagulation Laboratory Abnormalities (All Cycles) - Q3W Regimen
Description: Participants who experienced coagulation laboratory test abnormalities were summarized according to worst toxicity grade observed for each coagulation laboratory test. Laboratory abnormalities were graded by NCI CTCAE version 4.03. This outcome measure calculated the number of participants with coagulation laboratory abnormalities that were shifted from <=Grade 2 at baseline to Grade 3 or above, including the following parameter: partial thromboplastin time.
Time Frame: From baseline to end of treatment (approximately 32 months).
Population: All participants enrolled in Q3W regimen who received at least 1 full or partial dose of study medication and had at least 1 observation of the given coagulation laboratory test.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 91 | 5
Participants | 0 | 0 | 0 | 0 | 1 | 0

9. Primary Outcome: Number of Participants With DLTs - Q2W Regimen
Description: A DLT was any of the following AEs in the first cycle of treatment (within 28 days of first dose or until participant received second infusion if there were treatment delayed) in the single agent dose escalation. (1)Hematologic: including Grade 4 neutropenia lasting >7 days; Febrile neutropenia; Grade >=3 neutropenic infection; Grade 4 thrombocytopenia; treatment delay >14 days because of hematologic AE; (2) Hepatic: including Grade>=3 serum bilirubin, hepatic transaminase or alkaline phosphatase; ALT or AST>=3.0 x ULN concurrent with elevation in bilirubin>=2.0 x ULN; (3) Grade >=3 non-hematologic, non-hepatic major organ toxicities; delayed by >2 weeks in receiving the next scheduled cycle due to persisting toxicities attributable to PF-06647020. Grade >=3 headache lasting >48 hours in presence of supportive care. A participant was on study for at least 28 days to be evaluable for DLT observation, and could be replaced if they terminated study participation earlier than 28 days.
Time Frame: First cycle, Day 1 up to Day 28
Population: All participants enrolled in Q2W regimen who received at least 1 dose of study medication and who did not have major treatment deviations during first cycle with a baseline disease assessment and at least 1 post baseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
Participants | 0 | 1 | 2

10. Primary Outcome: Number of Participants With Treatment-Emergent AEs - Q2W Regimen (All-Causality)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study medication.
Time Frame: From the time the participant took the first dose of study medication through the participant's last visit. (approximately 19 months)
Population: All participants enrolled in Q2W regimen who received at least 1 full or partial dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
Participants
  AEs | 3 | 10 | 12
  SAEs | 1 | 4 | 7

11. Primary Outcome: Number of Participants With Treatment-Emergent AEs - Q2W Regimen (Treatment-Related)
Description: as for outcome 3
Time Frame: as for outcome 10
Population: All participants enrolled in Q2W regimen who received at least 1 full or partial dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
Participants
  AEs | 3 | 10 | 12
  SAEs | 0 | 2 | 2

12. Primary Outcome: Number of Participants With Treatment-Emergent AEs Categorized by Seriousness - Q2W Regimen (All-Causality and Treatment-Related)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study medication. All AEs were graded by the investigator according to the NCI CTCAE version 4.03. Grade 1 AEs are mild AEs; Grade 2 AEs are moderate AEs; Grade 3 AEs are severe AEs, Grade 4 AEs are life-threatening consequences and Grade 5 AEs are deaths related to AEs. Each AE was counted once for the participant in the most severe severity.
Time Frame: as for outcome 10
Population: All participants enrolled in Q2W regimen who received at least 1 full or partial dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
Participants
  Grade 1 (all-causality) | 0 | 0 | 0
  Grade 2 (all-causality) | 2 | 3 | 2
  Grade 3 (all-causality) | 1 | 5 | 7
  Grade 4 (all-causality) | 0 | 2 | 2
  Grade 5 (all-causality) | 0 | 0 | 1
  Missing or Unknown (all-causality) | 0 | 0 | 0
  Grade 1 (treatment-related) | 0 | 0 | 0
  Grade 2 (treatment-related) | 3 | 4 | 5
  Grade 3 (treatment-related) | 0 | 4 | 6
  Grade 4 (treatment-related) | 0 | 2 | 1
  Grade 5 (treatment-related) | 0 | 0 | 0
  Missing or Unknown (treatment-related) | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Hematology Laboratory Abnormalities (All Cycles) - Q2W Regimen
Description: Participants who experienced hematology laboratory test abnormalities were summarized according to worst toxicity grade observed for each hematology laboratory test. Laboratory abnormalities were graded by NCI CTCAE version 4.03. This outcome measure calculated the number of participants with hematology laboratory abnormalities that were shifted from <=Grade 2 at baseline to Grade 3 or above, including the following parameters: absolute neutrophils, lymphopenia, white blood cell, anemia.
Time Frame: From baseline to end of treatment (approximately 19 months).
Population: All participants enrolled in Q2W regimen who received at least 1 full or partial dose of study medication and had at least 1 observation of the given hematology laboratory test.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
Participants
  Absolute neutrophils | 0 | 3 | 5
  Lymphopenia | 0 | 0 | 4
  White blood cells | 0 | 2 | 2
  Anemia | 0 | 0 | 1

14. Primary Outcome: Number of Participants With Chemistry Laboratory Abnormalities (All Cycles) - Q2W Regimen
Description: Participants who experienced chemistry laboratory test abnormalities were summarized according to worst toxicity grade observed for each chemistry laboratory test. Laboratory abnormalities were graded by NCI CTCAE version 4.03. This outcome measure calculated the number of participants with chemistry laboratory abnormalities that were shifted from <=Grade 2 at baseline to Grade 3 or above, including the following parameters: hypokalemia, hyponatremia, hypomagnesemia, hypoalbuminemia, hypocalcemia, hypophosphatemia, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase.
Time Frame: From baseline to end of treatment (approximately 19 months).
Population: All participants enrolled in Q2W regimen who received at least 1 full or partial dose of study medication and had at least 1 observation of the given chemistry laboratory test.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
Participants
  Hypokalemia | 0 | 1 | 2
  Hyponatremia | 0 | 1 | 2
  Hypomagnesemia | 0 | 0 | 2
  Hypoalbuminemia | 0 | 1 | 1
  Hypocalcemia | 1 | 0 | 1
  Hypophosphatemia | 0 | 1 | 0
  Alanine aminotransferase | 0 | 0 | 1
  Aspartate aminotransferase | 0 | 0 | 1
  Alkaline phosphatase | 0 | 0 | 1

15. Primary Outcome: Number of Participants With Urinalysis Laboratory Abnormalities (All Cycles) - Q2W Regimen
Description: as for outcome 7
Time Frame: Baseline and Day 1 of Cycle 1
Population: All participants enrolled in Q2W regimen who received at least 1 full or partial dose of study medication and had at least 1 observation of the given urinalysis laboratory test.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 0 | 2 | 1
Participants | 0 | 0 | 0

16. Primary Outcome: Number of Participants With Coagulation Laboratory Abnormalities (All Cycles) - Q2W Regimen
Description: Participants who experienced coagulation laboratory test abnormalities were summarized according to worst toxicity grade observed for each urinalysis laboratory test. Laboratory abnormalities were graded by NCI CTCAE version 4.03. This outcome measure calculated the number of participants with coagulation laboratory abnormalities that were shifted from <=Grade 2 at baseline to Grade 3 or above, including the following parameter: prothrombin time international normalized ratio.
Time Frame: From baseline to end of treatment (approximately 19 months).
Population: All participants enrolled in Q2W regimen who received at least 1 full or partial dose of study medication and had at least 1 observation of the given coagulation laboratory test.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
Participants | 0 | 0 | 1

17. Secondary Outcome: Area Under the Concentration-Time Profile From Time 0 to Time Tau (AUCtau) for PF-06647020 - Q3W Regimen
Description: Tau refers to the dosing interval and it equals to 504 hours for the Q3W dosing. AUCtau is the area under the concentration-time profile from time 0 to time tau. AUCtau for PF-06647020 was determined using linear/log trapezoidal method.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: All participants enrolled in Q3W regimen (except DDI sub-study) who received at least 1 dose of study treatment and had sufficient information to estimate at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram•hour/milliliter (µg•hr/mL)
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
microgram•hour/milliliter (µg•hr/mL)
  Cycle 1, Single Dose: number analyzed (Participants) | 2 | 2 | 2 | 4 | 83 | 5
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4570 (30) | 4782 (61) | 6929 (80)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 41 | 2
  Cycle 4, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4201 (95) | 5834 (60) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

18. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for PF-06647020 -Q3W Regimen
Description: Cmax is maximum observed serum concentration. Cmax for PF-06647020 was observed directly from data.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (µg/mL)
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
microgram/milliliter (µg/mL)
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 65.77 (25) | 79.77 (45) | 96.11 (47)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 42 | 2
  Cycle 4, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 55.41 (53) | 92.94 (50) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

19. Secondary Outcome: Clearance (CL) for PF-06647020 - Q3W Regimen
Description: Clearance (CL) is a quantitative measure of the rate at which a drug substance is removed from the body. Clearance for PF-06647020 was calculated as dose/AUCinf for single dose and dose/AUCtau for multiple dose, where AUCinf was the area under the serum concentration-time profile from time 0 extrapolated to infinite time and AUCtau was the area under the concentration-time profile from time 0 to time tau (tau equals to 504 hours for the Q3W dosing).
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/hr)
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
Liter/hour (L/hr)
  Cycle 1, Single Dose: number analyzed (Participants) | 2 | 1 | 2 | 4 | 82 | 5
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 0.03464 (27) | 0.03956 (60) | 0.03694 (72)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 41 | 2
  Cycle 4, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 0.03640 (42) | 0.03121 (60) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

20. Secondary Outcome: Volume of Distribution at Steady State (Vss) for PF-06647020 - Q3W Regimen
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
Liter (L)
  Cycle 1, Single Dose: number analyzed (Participants) | 2 | 1 | 2 | 4 | 82 | 5
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 3.498 (26) | 3.199 (40) | 3.947 (52)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 37 | 2
  Cycle 4, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 3.230 (46) | 2.808 (47) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

21. Secondary Outcome: Terminal Half-Life (t1/2) for PF-06647020 - Q3W Regimen
Description: Terminal half-life (t1/2) is the time measured for the plasma concentration of drug to decrease by one half.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: day
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
day
  Cycle 1, Single Dose: number analyzed (Participants) | 2 | 1 | 2 | 4 | 82 | 5
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 3.600 (0.487) | 3.107 (1.161) | 3.514 (0.696)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 37 | 2
  Cycle 4, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4.013 (2.891) | 4.007 (1.496) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

22. Secondary Outcome: Observed Accumulation Ratio (Rac) for PF-06647020 - Q3W Regimen
Description: Rac is defined as observed accumulation ratio based on dose normalized AUCtau (AUCtau[dn]), where AUCtau is the area under the concentration-time profile from time 0 to time tau (tau equals to 504 hours for the Q3W dosing). Rac=Cycle 4 Day 1 AUCtau(dn) (multiple dose) /Cycle 1 Day 1 AUCtau(dn) (single Dose).
Time Frame: pre-dose, 1, 4 hours post-dose on Day 1 of Cycle 1 and Day 1 of Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 1 | 0 | 1 | 3 | 41 | 2
Ratio | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 1.046 (61) | 1.094 (39) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

23. Secondary Outcome: Time for Cmax (Tmax) for PF-06647020 - Q3W Regimen
Description: Tmax is the time for Cmax. Tmax for PF-06647020 was observed directly from data as time of first occurrence.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
hour
  Cycle 1, Single Dose | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 2.48 [0.950 to 4.17] | 1.08 [0.950 to 70.3] | 2.49 [0.983 to 24.1]
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 42 | 2
  Cycle 4, Multiple Dose | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 3.05 [0.967 to 24.0] | 1.65 [0.917 to 48.2] | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

24. Secondary Outcome: Area Under the Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) for PF-06647020 - Q3W Regimen
Description: AUClast is the area under the serum concentration-time profile from time 0 to the time of the last quantifiable concentration. AUClast for PF-06647020 was determined using linear/log trapezoidal method.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
µg•hr/mL
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4570 (30) | 4674 (63) | 4450 (198)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 42 | 2
  Cycle 4, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4157 (98) | 5428 (83) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

25. Secondary Outcome: Area Under the Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) for PF-06647020 - Q3W Regimen
Description: AUCinf is the area under the serum concentration-time profile from time 0 extrapolated to infinite time. AUCinf for PF-06647020 was calculated as AUClast + (Clast*/kel), where AUClast was the area under the serum concentration-time profile from time 0 to the time of the last quantifiable concentration, Clast* was the predicted serum concentration at the last quantifiable time point estimated from the log-linear regression analysis. kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
µg•hr/mL
  Cycle 1, Single Dose: number analyzed (Participants) | 2 | 1 | 2 | 4 | 82 | 5
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4637 (30) | 4829 (63) | 7052 (81)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 37 | 2
  Cycle 4, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4312 (102) | 6086 (62) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

26. Secondary Outcome: AUCtau for PF-06380101 - Q3W Regimen
Description: Tau refers to the dosing interval and it equals to 504 hours for the Q3W dosing. AUCtau is the area under the concentration-time profile from time 0 to time tau. AUCtau for PF-06380101 was determined using linear/log trapezoidal method.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram•hour/milliliter (ng•hr/mL)
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
nanogram•hour/milliliter (ng•hr/mL)
  Cycle 1, Single Dose: number analyzed (Participants) | 2 | 2 | 2 | 4 | 82 | 5
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 844.6 (46) | 803.9 (68) | 1022 (78)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 42 | 2
  Cycle 4, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 418.3 (106) | 647.9 (46) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

27. Secondary Outcome: Cmax for PF-06380101 - Q3W Regimen
Description: Cmax is maximum observed serum concentration. Cmax for PF-06380101 was observed directly from data.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
nanogram/milliliter (ng/mL)
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 7.156 (39) | 6.934 (69) | 7.660 (47)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 42 | 2
  Cycle 4, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 3.379 (84) | 5.746 (60) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

28. Secondary Outcome: t1/2 for PF-06380101 - Q3W Regimen
Description: Terminal half-life (t1/2) is the time measured for the plasma concentration of drug to decrease by one half.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: day
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
day
  Cycle 1, Single Dose: number analyzed (Participants) | 1 | 1 | 2 | 4 | 81 | 4
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 3.150 (0.426) | 2.881 (0.604) | 3.210 (0.473)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 40 | 2
  Cycle 4, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 2.827 (0.391) | 2.781 (0.676) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

29. Secondary Outcome: Rac for PF-06380101 - Q3W Regimen
Description: as for outcome 22
Time Frame: pre-dose, 1, 4 hours post-dose on Day 1 of Cycle 1 and Day 1 of Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 1 | 0 | 1 | 3 | 42 | 2
Ratio | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 0.5454 (40) | 0.8916 (41) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

30. Secondary Outcome: Tmax for PF-06380101 - Q3W Regimen
Description: Tmax is the time for Cmax. Tmax for PF-06380101 was observed directly from data as time of first occurrence.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
hour
  Cycle 1, Single Dose | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 23.6 [4.00 to 48.0] | 23.9 [3.90 to 141] | 23.4 [4.00 to 74.0]
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 42 | 2
  Cycle 4, Multiple Dose | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 23.8 [23.6 to 24.0] | 21.9 [3.67 to 96.0] | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

31. Secondary Outcome: AUClast for PF-06380101 - Q3W Regimen
Description: AUClast is the area under the serum concentration-time profile from time 0 to the time of the last quantifiable concentration. AUClast for PF-06380101 was determined using linear/log trapezoidal method.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
ng•hr/mL
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 844.6 (46) | 799.3 (68) | 490.5 (615)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 42 | 2
  Cycle 4, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 418.5 (106) | 643.6 (48) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

32. Secondary Outcome: AUCinf for PF-06380101 - Q3W Regimen
Description: AUCinf is the area under the serum concentration-time profile from time 0 extrapolated to infinite time. AUCinf for PF-06380101 was calculated as AUClast + (Clast*/kel), where AUClast was the area under the serum concentration-time profile from time 0 to the time of the last quantifiable concentration, Clast* was the predicted serum concentration at the last quantifiable time point estimated from the log-linear regression analysis. kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
ng•hr/mL
  Cycle 1, Single Dose: number analyzed (Participants) | 1 | 1 | 2 | 4 | 81 | 4
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 851.4 (45) | 812.2 (68) | 1020 (95)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 40 | 2
  Cycle 4, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 422.9 (105) | 645.2 (48) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

33. Secondary Outcome: AUCtau for hu6M024 mAb - Q3W Regimen
Description: Tau refers to the dosing interval and it equals to 504 hours for the Q3W dosing. AUCtau is the area under the concentration-time profile from time 0 to time tau. AUCtau for hu6M024 mAb was determined using linear/log trapezoidal method.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
µg•hr/mL
  Cycle 1, Single Dose: number analyzed (Participants) | 2 | 2 | 2 | 4 | 83 | 5
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 6968 (32) | 5562 (62) | 8451 (78)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 41 | 2
  Cycle 4, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 6122 (145) | 6210 (80) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

34. Secondary Outcome: Cmax for hu6M024 mAb - Q3W Regimen
Description: Cmax is maximum observed serum concentration. Cmax for hu6M024 mAb was observed directly from data.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
µg/mL
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 83.33 (20) | 84.83 (43) | 99.37 (47)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 42 | 2
  Cycle 4, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 77.76 (76) | 82.33 (40) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

35. Secondary Outcome: t1/2 for hu6M024 mAb - Q3W Regimen
Description: Terminal half-life (t1/2) is the time measured for the plasma concentration of drug to decrease by one half.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: day
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
day
  Cycle 1, Single Dose: number analyzed (Participants) | 2 | 2 | 2 | 4 | 81 | 5
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4.505 (0.650) | 3.674 (1.512) | 4.386 (0.895)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 0 | 0 | 1 | 3 | 37 | 2
  Cycle 4, Multiple Dose |  |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 5.087 (2.626) | 5.232 (2.259) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

36. Secondary Outcome: Rac for hu6M024 mAb - Q3W Regimen
Description: as for outcome 22
Time Frame: pre-dose, 1, 4 hours post-dose on Day 1 of Cycle 1 and Day 1 of Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 1 | 0 | 1 | 3 | 41 | 2
Ratio | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 1.022 (108) | 0.9865 (48) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

37. Secondary Outcome: Tmax for hu6M024 mAb - Q3W Regimen
Description: Tmax is the time for Cmax. Tmax for hu6M024 mAb was observed directly from data as time of first occurrence.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
hour
  Cycle 1, Single Dose | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4.00 [0.950 to 4.17] | 3.70 [0.933 to 24.1] | 2.31 [0.983 to 4.00]
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 42 | 2
  Cycle 4, Multiple Dose | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 3.05 [1.00 to 23.6] | 3.90 [1.00 to 41.8] | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

38. Secondary Outcome: AUClast for hu6M024 mAb - Q3W Regimen
Description: AUClast is the area under the serum concentration-time profile from time 0 to the time of the last quantifiable concentration. AUClast for hu6M024 mAb was determined using linear/log trapezoidal method.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
µg•hr/mL
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 6969 (32) | 5449 (64) | 5247 (221)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 1 | 0 | 1 | 3 | 42 | 2
  Cycle 4, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 6127 (147) | 5885 (97) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

39. Secondary Outcome: AUCinf for hu6M024 mAb - Q3W Regimen
Description: AUCinf is the area under the serum concentration-time profile from time 0 extrapolated to infinite time. AUCinf for hu6M024 mAb was calculated as AUClast + (Clast*/kel), where AUClast was the area under the serum concentration-time profile from time 0 to the time of the last quantifiable concentration, Clast* was the predicted serum concentration at the last quantifiable time point estimated from the log-linear regression analysis. kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 4 (21 days cycle).
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 85 | 6
µg•hr/mL
  Cycle 1, Single Dose: number analyzed (Participants) | 2 | 2 | 2 | 4 | 81 | 5
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 7189 (32) | 5608 (65) | 8760 (80)
  Cycle 4, Multiple Dose: number analyzed (Participants) | 0 | 0 | 1 | 3 | 37 | 2
  Cycle 4, Multiple Dose |  |  | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 6517 (156) | 6191 (94) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated.

40. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) and Neutralizing Antibody (NAb) of PF-06647020 - Q3W Regimen
Description: To evaluate the immunogenicity as measured by presence of ADA and NAb in participants treated with PF-06647020.
Time Frame: Prior to the start of treatment on Day 1 of Cycle 1 up to end of treatment (approximately 31 months).
Population: All participants enrolled in Q3W regimen who received at least 1 dose of study treatment and had at least 1 ADA sample collected.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 0.2 mg/kg（Q3W Regimen） | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen)
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 96 | 6
Participants
  Overall incidence of ADA: number analyzed (Participants) | 2 | 2 | 2 | 4 | 93 | 5
  Overall incidence of ADA | 1 | 0 | 0 | 0 | 10 | 0
  Overall incidence of NAb: number analyzed (Participants) | 2 | 2 | 2 | 4 | 93 | 5
  Overall incidence of NAb | 1 | 0 | 0 | 0 | 9 | 0

41. Secondary Outcome: Percentage of Participants With Objective Response - Q3W Regimen
Description: Percentage of participants with objective response based on assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline, every 6 weeks from the start of treatment until disease progression, death or withdrawal from treatment (approximately 32 months).
Population: Participants enrolled in Q3W regimen with measurable disease (non-small cell lung cancer [NSCLC], ovarian cancer [OVCA], triple negative breast cancer [TNBC]) who had received at least 1 dose of study medication and had a baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- NSCLC - Q3W Regimen: Participants with NSCLC received PF-06647020 on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
- OVCA - Q3W Regimen: Participants with OVCA received PF-06647020 on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
- TNBC - Q3W Regimen: Participants with TNBC received PF-06647020 on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
Arm/Group | NSCLC - Q3W Regimen | OVCA - Q3W Regimen | TNBC - Q3W Regimen
Number analyzed (Participants) | 25 | 44 | 29
Percentage of participants | 16.0 [4.5 to 36.1] | 27.3 [15.0 to 42.8] | 20.7 [8.0 to 39.7]

42. Secondary Outcome: Duration of Response - Q3W Regimen
Description: Duration of response (DoR) was the time from first documentation of PR or CR to date of first documentation of progressive disease (PD) or death due to any cause. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. PD was defined as at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of one or more new lesions.
Time Frame: as for outcome 41
Population: Participants enrolled in Q3W regimen with measurable disease (NSCLC, OVCA, TNBC) who had received at least 1 dose of study medication and had a baseline tumor assessment. DoR was only for the subset participants with an objective response.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | NSCLC - Q3W Regimen | OVCA - Q3W Regimen | TNBC - Q3W Regimen
Number analyzed (Participants) | 4 | 12 | 6
month | 5.7 [1.5 to 9.9] | 4.2 [2.8 to 8.3] | 4.3 [1.3 to 10.2]

43. Secondary Outcome: Disease Control Rate - Q3W Regimen
Description: The disease control rate (DCR) was defined as the percentage of participants with a confirmed CR, PR, non-CR/non-PD or stable disease (SD) according to the appropriate analysis set. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 41
Population: Participants enrolled in Q3W regimen with measurable disease (NSCLC, OVCA, TNBC) who had received at least 1 dose of study medication and had a baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NSCLC - Q3W Regimen | OVCA - Q3W Regimen | TNBC - Q3W Regimen
Number analyzed (Participants) | 25 | 44 | 29
Percentage of participants | 56.0 [34.93 to 75.60] | 72.7 [57.21 to 85.04] | 48.3 [29.45 to 67.47]

44. Secondary Outcome: Time to Progression - Q3W Regimen
Description: Time to progression (TTP) was the time from start date to the date of the first documentation of PD. PD was defined as at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of one or more new lesions.
Time Frame: as for outcome 41
Population: as for outcome 43
Measure: Median (95% Confidence Interval); unit: month
Groups:
- NSCLC - Q3W Regimen: Participants with NSCL received PF-06647020 on Day 1 of each 21-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
Arm/Group | NSCLC - Q3W Regimen | OVCA - Q3W Regimen | TNBC - Q3W Regimen
Number analyzed (Participants) | 25 | 44 | 29
month | 2.9 [1.4 to 6.1] | 3.1 [2.3 to 5.5] | 2.2 [1.4 to 5.5]

45. Secondary Outcome: Progression Free Survival - Q3W Regimen
Description: Progression free survival (PFS) was the time from randomization date to date of first documentation of PD or death due to any cause. PD was defined as at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of one or more new lesions.
Time Frame: as for outcome 41
Population: as for outcome 43
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | NSCLC - Q3W Regimen | OVCA - Q3W Regimen | TNBC - Q3W Regimen
Number analyzed (Participants) | 25 | 44 | 29
month | 2.9 [1.4 to 6.1] | 2.9 [2.3 to 5.5] | 1.5 [1.4 to 4.3]

46. Secondary Outcome: Dose Normalized AUCinf [AUCinf(dn)] for PF-06647020 [DDI Sub-Study]
Description: AUCinf is the area under the serum concentration-time profile from time 0 extrapolated to infinite time. AUCinf(dn) was defined as dose normalized AUCinf and calculated as AUCinf/dose.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 2 (21 days cycle).
Population: The drug-drug interaction (DDI) sub-study was determined to evaluate the effect of multiple dose fluconazole on the PK of PF-06380101 (payload), when fluconazole was co-administered with PF-06647020. The analysis population included participants who participated in the DDI sub-study, and had at least one of the study required PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL/mg
Groups:
- PF-06647020 2.8 mg/kg (Q3W-DDI): Participants who participated in the DDI sub-study received a single-dose of PF-06647020 intravenously at 2.8 mg/kg on Cycle 1 Day 1 (Period A).
- PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI): Participants who participated in the DDI sub-study received a single dose of PF-06647020 intravenously at 1.4 mg/kg on Cycle 2 Day 1 (Period B), in combination with fluconazole. Participants started with a loading dose of 400 mg fluconazole by mouth (PO) on the morning of Cycle 1 Day 21 and continued to take fluconazole in the morning at 200 mg PO daily from Cycle 2 Day 1 through Cycle 2 Day 7.
Arm/Group | PF-06647020 2.8 mg/kg (Q3W-DDI) | PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI)
Number analyzed (Participants) | 10 | 8
µg•hr/mL/mg | 29.56 (46) | 23.47 (53)
Statistical Analysis 1: Comparison: PF-06647020 2.8 mg/kg (Q3W-DDI) vs PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI); Test: PF-06647020 1.4 mg/kg + Fluconazole(Q3W-DDI) group; Reference: PF-06647020 2.8 mg/kg (Q3W-DDI) group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; p = 0.3105, ANOVA; Geometric Mean Ratio (GMR) = 79.38, 90% CI 2-sided [54.01 to 116.65]

47. Secondary Outcome: Dose Normalized AUClast [AUClast(dn)] for PF-06647020 [DDI Sub-Study]
Description: AUClast is the area under the serum concentration-time profile from time 0 to the time of the last quantifiable concentration. AUClast(dn) was defined as dose normalized AUClast and calculated as AUClast/dose.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 2 (21 days cycle).
Population: Participants who participated in the DDI sub-study, and had at least one of the study required PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL/mg
Arm/Group | PF-06647020 2.8 mg/kg (Q3W-DDI) | PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI)
Number analyzed (Participants) | 11 | 10
µg•hr/mL/mg | 31.51 (51) | 24.34 (50)
Statistical Analysis 1: Comparison: PF-06647020 2.8 mg/kg (Q3W-DDI) vs PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI); Test: PF-06647020 1.4 mg/kg + Fluconazole(Q3W-DDI) group; Reference: PF-06647020 2.8 mg/kg (Q3W-DDI) group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; p = 0.2316, ANOVA; Geometric Mean Ratio (GMR) = 77.23, 90% CI 2-sided [53.80 to 110.87]

48. Secondary Outcome: Dose Normalized AUCtau [AUCtau(dn)] for PF-06647020 [DDI Sub-Study]
Description: AUCtau is the area under the concentration-time profile from time 0 to time tau. AUCtau(dn) was defined as dose normalized AUCtau and calculated as AUCtau/dose.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 2 (21 days cycle).
Population: Participants who participated in the DDI sub-study, and had at least one of the study required PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL/mg
Arm/Group | PF-06647020 2.8 mg/kg (Q3W-DDI) | PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI)
Number analyzed (Participants) | 10 | 10
µg•hr/mL/mg | 29.25 (46) | 24.85 (48)
Statistical Analysis 1: Comparison: PF-06647020 2.8 mg/kg (Q3W-DDI) vs PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI); Test: PF-06647020 1.4 mg/kg + Fluconazole(Q3W-DDI) group; Reference: PF-06647020 2.8 mg/kg (Q3W-DDI) group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; p = 0.4264, ANOVA; Geometric Mean Ratio (GMR) = 84.97, 90% CI 2-sided [60.05 to 120.22]

49. Secondary Outcome: Dose Normalized Cmax [Cmax(dn)] for PF-06647020 [DDI Sub-Study]
Description: Cmax is maximum observed serum concentration. Cmax(dn) was defined as dose normalized Cmax and calculated as Cmax/dose.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 2 (21 days cycle).
Population: Participants who participated in the DDI sub-study, and had at least one of the study required PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL/mg
Arm/Group | PF-06647020 2.8 mg/kg (Q3W-DDI) | PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI)
Number analyzed (Participants) | 11 | 10
µg/mL/mg | 0.5010 (49) | 0.4425 (39)
Statistical Analysis 1: Comparison: PF-06647020 2.8 mg/kg (Q3W-DDI) vs PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI); Test: PF-06647020 1.4 mg/kg + Fluconazole(Q3W-DDI) group; Reference: PF-06647020 2.8 mg/kg (Q3W-DDI) group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; p = 0.5123, ANOVA; Geometric Mean Ratio (GMR) = 88.32, 90% CI 2-sided [64.03 to 121.82]

50. Secondary Outcome: AUCinf(dn) for PF-06380101 [DDI Sub-Study]
Description: as for outcome 46
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 2 (21 days cycle).
Population: Participants who participated in the DDI sub-study, and had at least one of the study required PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL/mg
Arm/Group | PF-06647020 2.8 mg/kg (Q3W-DDI) | PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI)
Number analyzed (Participants) | 11 | 10
ng•hr/mL/mg | 5.787 (116) | 5.275 (123)
Statistical Analysis 1: Comparison: PF-06647020 2.8 mg/kg (Q3W-DDI) vs PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI); Test: PF-06647020 1.4 mg/kg + Fluconazole(Q3W-DDI) group; Reference: PF-06647020 2.8 mg/kg (Q3W-DDI) group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; p = 0.8240, ANOVA; Geometric Mean Ratio (GMR) = 91.15, 90% CI 2-sided [44.79 to 185.50]

51. Secondary Outcome: AUClast(dn) for PF-06380101 [DDI Sub-Study]
Description: as for outcome 47
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 2 (21 days cycle).
Population: Participants who participated in the DDI sub-study, and had at least one of the study required PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL/mg
Arm/Group | PF-06647020 2.8 mg/kg (Q3W-DDI) | PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI)
Number analyzed (Participants) | 11 | 10
ng•hr/mL/mg | 5.681 (112) | 5.089 (128)
Statistical Analysis 1: Comparison: PF-06647020 2.8 mg/kg (Q3W-DDI) vs PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI); Test: PF-06647020 1.4 mg/kg + Fluconazole(Q3W-DDI) group; Reference: PF-06647020 2.8 mg/kg (Q3W-DDI) group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; p = 0.7922, ANOVA; Geometric Mean Ratio (GMR) = 89.58, 90% CI 2-sided [43.94 to 182.62]

52. Secondary Outcome: AUCtau(dn) for PF-06380101 [DDI Sub-Study]
Description: as for outcome 48
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 2 (21 days cycle).
Population: Participants who participated in the DDI sub-study, and had at least one of the study required PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL/mg
Arm/Group | PF-06647020 2.8 mg/kg (Q3W-DDI) | PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI)
Number analyzed (Participants) | 11 | 10
ng•hr/mL/mg | 5.746 (115) | 5.239 (123)
Statistical Analysis 1: Comparison: PF-06647020 2.8 mg/kg (Q3W-DDI) vs PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI); Test: PF-06647020 1.4 mg/kg + Fluconazole(Q3W-DDI) group; Reference: PF-06647020 2.8 mg/kg (Q3W-DDI) group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; p = 0.8240, ANOVA; Geometric Mean Ratio (GMR) = 91.17, 90% CI 2-sided [44.87 to 185.25]

53. Secondary Outcome: Cmax(dn) for PF-06380101 [DDI Sub-Study]
Description: Cmax is maximum observed serum concentration. Cmax(dn) was defined as dose normalized Cmax and calculated as Cmax/dose.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 2 (21 days cycle).
Population: Participants who participated in the DDI sub-study, and had at least one of the study required PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | PF-06647020 2.8 mg/kg (Q3W-DDI) | PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI)
Number analyzed (Participants) | 11 | 10
ng/mL/mg | 0.04336 (113) | 0.04436 (118)
Statistical Analysis 1: Comparison: PF-06647020 2.8 mg/kg (Q3W-DDI) vs PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI); Test: PF-06647020 1.4 mg/kg + Fluconazole(Q3W-DDI) group; Reference: PF-06647020 2.8 mg/kg (Q3W-DDI) group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; p = 0.9553, ANOVA; Geometric Mean Ratio (GMR) = 102.31, 90% CI 2-sided [51.08 to 204.90]

54. Secondary Outcome: AUCinf(dn) for hu6M024 mAb [DDI Sub-Study]
Description: as for outcome 46
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 2 (21 days cycle).
Population: Participants who participated in the DDI sub-study, and had at least one of the study required PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL/mg
Arm/Group | PF-06647020 2.8 mg/kg (Q3W-DDI) | PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI)
Number analyzed (Participants) | 11 | 9
µg•hr/mL/mg | 31.94 (45) | 25.92 (46)
Statistical Analysis 1: Comparison: PF-06647020 2.8 mg/kg (Q3W-DDI) vs PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI); Test: PF-06647020 1.4 mg/kg + Fluconazole(Q3W-DDI) group; Reference: PF-06647020 2.8 mg/kg (Q3W-DDI) group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; p = 0.2951, ANOVA; Geometric Mean Ratio (GMR) = 81.14, 90% CI 2-sided [57.99 to 113.54]

55. Secondary Outcome: AUClast(dn) for hu6M024 mAb [DDI Sub-Study]
Description: as for outcome 47
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 2 (21 days cycle).
Population: Participants who participated in the DDI sub-study, and had at least one of the study required PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL/mg
Arm/Group | PF-06647020 2.8 mg/kg (Q3W-DDI) | PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI)
Number analyzed (Participants) | 11 | 10
µg•hr/mL/mg | 31.30 (44) | 26.30 (48)
Statistical Analysis 1: Comparison: PF-06647020 2.8 mg/kg (Q3W-DDI) vs PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI); Test: PF-06647020 1.4 mg/kg + Fluconazole(Q3W-DDI) group; Reference: PF-06647020 2.8 mg/kg (Q3W-DDI) group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; p = 0.3769, ANOVA; Geometric Mean Ratio (GMR) = 84.02, 90% CI 2-sided [60.24 to 117.19]

56. Secondary Outcome: AUCtau(dn) for hu6M024 mAb [DDI Sub-Study]
Description: as for outcome 48
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 2 (21 days cycle).
Population: Participants who participated in the DDI sub-study, and had at least one of the study required PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL/mg
Arm/Group | PF-06647020 2.8 mg/kg (Q3W-DDI) | PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI)
Number analyzed (Participants) | 11 | 10
µg•hr/mL/mg | 31.29 (44) | 26.96 (46)
Statistical Analysis 1: Comparison: PF-06647020 2.8 mg/kg (Q3W-DDI) vs PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI); Test: PF-06647020 1.4 mg/kg + Fluconazole(Q3W-DDI) group; Reference: PF-06647020 2.8 mg/kg (Q3W-DDI) group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; p = 0.4385, ANOVA; Geometric Mean Ratio (GMR) = 86.15, 90% CI 2-sided [62.20 to 119.32]

57. Secondary Outcome: Cmax(dn) for hu6M024 mAb [DDI Sub-Study]
Description: Cmax is maximum observed serum concentration. Cmax(dn) was defined as dose normalized Cmax and calculated as Cmax/dose.
Time Frame: pre-dose, 1, 4, 24, 72, 168, 336 hours post-dose for Cycle 1 and Cycle 2 (21 days cycle).
Population: Participants who participated in the DDI sub-study, and had at least one of the study required PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL/mg
Arm/Group | PF-06647020 2.8 mg/kg (Q3W-DDI) | PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI)
Number analyzed (Participants) | 11 | 10
µg/mL/mg | 0.4378 (59) | 0.3885 (37)
Statistical Analysis 1: Comparison: PF-06647020 2.8 mg/kg (Q3W-DDI) vs PF-06647020 1.4 mg/kg + Fluconazole (Q3W-DDI); Test: PF-06647020 1.4 mg/kg + Fluconazole(Q3W-DDI) group; Reference: PF-06647020 2.8 mg/kg (Q3W-DDI) group; Test type: Other — The ratio and 90% confidence interval were expressed as percentages; p = 0.5678, ANOVA; Geometric Mean Ratio (GMR) = 88.75, 90% CI 2-sided [62.24 to 126.56]

58. Secondary Outcome: AUCtau for PF-06647020 - Q2W Regimen
Description: Tau refers to the dosing interval and it equals to 336 hours for the Q2W dosing. AUCtau is the area under the concentration-time profile from time 0 to time tau. AUCtau for PF-06647020 was determined using linear/log trapezoidal method.
Time Frame: pre-dose, end of infusion, 4, 24, 72, 168 hours post-dose, Day 15 (pre-dose, end of infusion) for Cycle 1 and Cycle 3 (28 days cycle).
Population: All participants enrolled in Q2W regimen who received at least 1 dose of study treatment and had sufficient information to estimate at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
µg•hr/mL
  Cycle 1, Single Dose | 3627 (62) | 6541 (38) | 6319 (45)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 9858 (21) | 6933 (43)

59. Secondary Outcome: Cmax for PF-06647020 -Q2W Regimen
Description: Cmax is maximum observed serum concentration. Cmax for PF-06647020 was observed directly from data.
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
µg/mL
  Cycle 1, Single Dose | 97.79 (14) | 99.69 (32) | 90.28 (32)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 114.7 (26) | 81.91 (34)

60. Secondary Outcome: Vss for PF-06647020 - Q2W Regimen
Description: as for outcome 20
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
Liter
  Cycle 1, Single Dose: number analyzed (Participants) | 2 | 9 | 12
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 2.566 (44) | 2.953 (36)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 2.349 (24) | 3.106 (32)

61. Secondary Outcome: CL for PF-06647020 - Q2W Regimen
Description: Clearance (CL) is a quantitative measure of the rate at which a drug substance is removed from the body. Clearance for PF-06647020 was calculated as dose/AUCinf for single dose and dose/AUCtau for multiple dose, where AUCinf was the area under the serum concentration-time profile from time 0 extrapolated to infinite time and AUCtau was the area under the concentration-time profile from time 0 to time tau (tau equals to 336 hours for the Q2W dosing).
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
L/hr
  Cycle 1, Single Dose: number analyzed (Participants) | 2 | 9 | 12
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 0.03075 (49) | 0.03238 (39)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 0.02044 (25) | 0.02688 (35)

62. Secondary Outcome: t1/2 for PF-06647020 - Q2W Regimen
Description: Terminal half-life (t1/2) is the time measured for the plasma concentration of drug to decrease by one half.
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: day
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
day
  Cycle 1, Single Dose: number analyzed (Participants) | 2 | 9 | 12
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 2.700 (0.625) | 2.874 (0.385)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 3.633 (0.415) | 3.600 (0.583)

63. Secondary Outcome: Rac for PF-06647020 - Q2W Regimen
Description: Rac is defined as observed accumulation ratio based on dose normalized AUCtau (AUCtau[dn]), where AUCtau is the area under the concentration-time profile from time 0 to time tau (tau equals to 336 hours for the Q2W dosing). Rac= Cycle 3 Day 1 AUCtau(dn) (multiple dose) /Cycle 1 Day 1 AUCtau(dn) (single Dose).
Time Frame: pre-dose, end of infusion, 4 hours post-dose on Day 1 of Cycle 1 and Day 1 of Cycle 3 (28 days cycle).
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 1 | 7 | 10
Ratio | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 1.425 (35) | 1.211 (18)

64. Secondary Outcome: Tmax for PF-06647020 - Q2W Regimen
Description: Tmax is the time for Cmax. Tmax for PF-06647020 was observed directly from data as time of first occurrence.
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
hour
  Cycle 1, Single Dose | 3.98 [0.983 to 4.02] | 2.45 [0.983 to 23.7] | 1.05 [0.900 to 4.00]
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 1.07 [0.983 to 23.9] | 2.36 [0.983 to 4.03]

65. Secondary Outcome: AUClast for PF-06647020 - Q2W Regimen
Description: as for outcome 24
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
µg•hr/mL
  Cycle 1, Single Dose | 3641 (62) | 6490 (39) | 6342 (46)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 9864 (20) | 7000 (43)

66. Secondary Outcome: AUCinf for PF-06647020 - Q2W Regimen
Description: AUCinf is the area under the serum concentration-time profile from time 0 extrapolated to infinite time. AUCinf was calculated as AUClast + (Clast*/kel), where AUClast was the area under the serum concentration-time profile from time 0 to the time of the last quantifiable concentration, Clast* was the predicted serum concentration at the last quantifiable time point estimated from the log-linear regression analysis. kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
µg•hr/mL
  Cycle 1, Single Dose: number analyzed (Participants) | 2 | 9 | 12
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 6798 (41) | 6535 (46)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 10570 (22) | 7445 (44)

67. Secondary Outcome: AUCtau for PF-06380101 - Q2W Regimen
Description: Tau refers to the dosing interval and it equals to 336 hours for the Q2W dosing. AUCtau is the area under the concentration-time profile from time 0 to time tau. AUCtau for PF-06380101 was determined using linear/log trapezoidal method.
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
ng•hr/mL
  Cycle 1, Single Dose | 568.9 (12) | 860.3 (52) | 740.5 (62)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 731.5 (61) | 589.8 (33)

68. Secondary Outcome: Cmax for PF-06380101 - Q2W Regimen
Description: Cmax is maximum observed serum concentration. Cmax for PF-06380101 was observed directly from data.
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
ng/mL
  Cycle 1, Single Dose | 6.084 (59) | 6.665 (49) | 5.779 (59)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4.857 (66) | 4.248 (34)

69. Secondary Outcome: t1/2 for PF-06380101 - Q2W Regimen
Description: Terminal half-life (t1/2) is the time measured for the plasma concentration of drug to decrease by one half.
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: day
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
day
  Cycle 1, Single Dose | 2.507 (0.411) | 2.646 (0.453) | 2.592 (0.331)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 6 | 10
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 2.755 (0.653) | 3.007 (0.373)

70. Secondary Outcome: Rac for PF-06380101 - Q2W Regimen
Description: as for outcome 63
Time Frame: pre-dose, end of infusion, 4 hours post-dose on Day 1 of Cycle 1 and Day 1 of Cycle 3 (28 days cycle).
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 1 | 7 | 10
Ratio | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 0.9980 (26) | 0.9657 (25)

71. Secondary Outcome: Tmax for PF-06380101 - Q2W Regimen
Description: Tmax is the time for Cmax. Tmax for PF-06380101 was observed directly from data as time of first occurrence.
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
hour
  Cycle 1, Single Dose | 3.98 [3.98 to 4.02] | 4.05 [3.75 to 72.1] | 24.7 [3.72 to 48.5]
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 71.7 [3.75 to 166] | 22.8 [3.75 to 48.3]

72. Secondary Outcome: AUClast for PF-06380101- Q2W Regimen
Description: as for outcome 31
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
ng•hr/mL
  Cycle 1, Single Dose | 569.9 (12) | 866.0 (53) | 743.5 (63)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 728.9 (60) | 593.3 (33)

73. Secondary Outcome: AUCinf for PF-06380101- Q2W Regimen
Description: as for outcome 66
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
ng•hr/mL
  Cycle 1, Single Dose | 584.4 (11) | 888.5 (54) | 763.2 (62)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 6 | 10
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 738.8 (69) | 617.9 (32)

74. Secondary Outcome: AUCtau for hu6M024 mAb- Q2W Regimen
Description: Tau refers to the dosing interval and it equals to 336 hours for the Q2W dosing. AUCtau is the area under the concentration-time profile from time 0 to time tau. AUCtau for hu6M024 mA was determined using linear/log trapezoidal method.
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
µg•hr/mL
  Cycle 1, Single Dose | 4089 (52) | 7325 (47) | 6911 (44)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 10440 (25) | 8432 (42)

75. Secondary Outcome: Cmax for hu6M024 mAb -Q2W Regimen
Description: Cmax is maximum observed serum concentration. Cmax for hu6M024 mAb was observed directly from data.
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
µg/mL
  Cycle 1, Single Dose | 72.04 (23) | 102.1 (38) | 86.26 (27)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 106.6 (37) | 89.66 (33)

76. Secondary Outcome: t1/2 for hu6M024 mAb - Q2W Regimen
Description: Terminal half-life (t1/2) is the time measured for the plasma concentration of drug to decrease by one half.
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: day
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
day
  Cycle 1, Single Dose: number analyzed (Participants) | 2 | 10 | 12
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 3.436 (0.750) | 3.645 (0.752)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 5 | 7
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 4.734 (0.670) | 4.124 (1.218)

77. Secondary Outcome: Rac for hu6M024 mAb - Q2W Regimen
Description: as for outcome 63
Time Frame: pre-dose, end of infusion, 4 hours post-dose on Day 1 of Cycle 1 and Day 1 of Cycle 3 (28 days cycle).
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 1 | 7 | 10
Ratio | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 1.280 (32) | 1.301 (35)

78. Secondary Outcome: Tmax for hu6M024 mAb - Q2W Regimen
Description: Tmax is the time for Cmax. Tmax for hu6M024 mAb was observed directly from data as time of first occurrence.
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Median (Full Range); unit: hour
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
hour
  Cycle 1, Single Dose | 3.98 [1.00 to 4.02] | 3.87 [0.983 to 4.35] | 1.05 [0.900 to 23.8]
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 1.05 [0.950 to 3.92] | 2.36 [0.983 to 24.1]

79. Secondary Outcome: AUClast for hu6M024 mAb - Q2W Regimen
Description: as for outcome 38
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
µg•hr/mL
  Cycle 1, Single Dose | 4103 (52) | 7368 (46) | 6949 (45)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 7 | 10
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 10460 (24) | 8555 (41)

80. Secondary Outcome: AUCinf for hu6M024 mAb - Q2W Regimen
Description: as for outcome 66
Time Frame: as for outcome 58
Population: as for outcome 58
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•hr/mL
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
µg•hr/mL
  Cycle 1, Single Dose: number analyzed (Participants) | 2 | 10 | 12
  Cycle 1, Single Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 7742 (47) | 7411 (48)
  Cycle 3, Multiple Dose: number analyzed (Participants) | 1 | 5 | 7
  Cycle 3, Multiple Dose | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 10950 (22) | 8275 (44)

81. Secondary Outcome: Number of Participants With ADA and NAb of PF-06647020 - Q2W Regimen
Description: To evaluate the immunogenicity as measured by presence of ADA and NAb in participants treated with PF-06647020.
Time Frame: 2 hours before the first dose up to 30 days after the last dose (approximately 18 months).
Population: All participants enrolled in Q2W regimen who received at least 1 dose of study treatment and had at least 1 ADA sample collected.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
Number analyzed (Participants) | 3 | 10 | 12
Participants
  Overall incidence of ADA | 1 | 0 | 0
  Overall incidence of NAb | 1 | 0 | 0

82. Secondary Outcome: Percentage of Participants With Objective Response - Q2W Regimen
Description: Percentage of participants with objective response based on assessment of CR or PR according to RECIST version 1.1. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline, every 8 weeks from the start of study treatment until disease progression, death or withdrawal from treatment (approximately 19 months).
Population: Participants enrolled in Q2W with measurable disease (NSCLC, OVCA) who had received at least 1 dose of study medication and had a baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- NSCLC - Q2W Regimen: Participants with NSCLC received PF-06647020 on Days 1 and 15 of each 28-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
- OVCA - Q2W Regimen: Participants with OVCA received PF-06647020 on Days 1 and 15 of each 28-day cycle as an IV infusion over approximately 60 minutes on an outpatient basis. Each participant received PF-06647020 until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
Arm/Group | NSCLC - Q2W Regimen | OVCA - Q2W Regimen
Number analyzed (Participants) | 6 | 19
Percentage of participants | 33.3 [4.3 to 77.7] | 26.3 [9.1 to 51.2]

83. Secondary Outcome: Duration of Response - Q2W Regimen
Description: For participants with an objective response, duration of response (DoR) was the time from first documentation of PR or CR to date of first documentation of PD or death due to any cause. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. PD was defined as at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of one or more new lesions.
Time Frame: as for outcome 82
Population: Participants enrolled in Q2W regimen with measurable disease (NSCLC, OVCA) who had received at least 1 dose of study medication and had a baseline tumor assessment. DoR was only for the subset participants with an objective response.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | NSCLC - Q2W Regimen | OVCA - Q2W Regimen
Number analyzed (Participants) | 2 | 5
month | NA [3.7 to NA] — NA indicates not calculable. Number of participants with confirmed objective response was too small to provide such summary statistics. | 6.5 [3.9 to 8.3]

84. Secondary Outcome: Disease Control Rate - Q2W Regimen
Description: The disease control rate (DCR) was defined as the percentage of participants with a confirmed CR, PR or SD according to the appropriate analysis set. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 82
Population: Participants enrolled in Q2W regimen with measurable disease (NSCLC, OVCA) who had received at least 1 dose of study medication and had a baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NSCLC - Q2W Regimen | OVCA - Q2W Regimen
Number analyzed (Participants) | 6 | 19
Percentage of participants | 50 [11.81 to 88.19] | 84.2 [60.42 to 96.62]

85. Secondary Outcome: Time to Progression - Q2W Regimen
Description: as for outcome 44
Time Frame: as for outcome 82
Population: as for outcome 84
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | NSCLC - Q2W Regimen | OVCA - Q2W Regimen
Number analyzed (Participants) | 6 | 19
month | 2.7 [1.0 to NA] — NA indicates not calculable. Number of participants with PD was too small to provide such summary statistics. | 3.8 [3.1 to 7.4]

86. Secondary Outcome: Progression Free Survival - Q2W Regimen
Description: as for outcome 45
Time Frame: as for outcome 82
Population: as for outcome 84
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | NSCLC - Q2W Regimen | OVCA - Q2W Regimen
Number analyzed (Participants) | 6 | 19
month | 2.7 [1.0 to NA] — NA indicates not calculable. Number of participants with PD or death was too small to provide such summary statistics. | 3.8 [3.1 to 7.4]

ADVERSE EVENTS:
Time Frame: From the time the participant took the first dose of study medication through the participant's last visit.(approximately 32 months)
Description: MedDRA 22.1 coding dictionary was applied for all AE tables. The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-06647020 0.2 mg/kg (Q3W Regimen) | PF-06647020 0.5 mg/kg (Q3W Regimen) | PF-06647020 1.25 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q3W Regimen) | PF-06647020 2.8 mg/kg (Q3W Regimen) | PF-06647020 3.7 mg/kg (Q3W Regimen) | PF-06647020 2.1 mg/kg (Q2W Regimen) | PF-06647020 2.8 mg/kg (Q2W Regimen) | PF-06647020 3.2 mg/kg (Q2W Regimen)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/4 | 13/96 | 0/6 | 0/3 | 0/10 | 2/12
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 1/4 | 33/96 | 2/6 | 1/3 | 4/10 | 7/12
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 4/4 | 93/96 | 6/6 | 3/3 | 10/10 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06647020 0.2 mg/kg (Q3W Regimen) (N=2) | PF-06647020 0.5 mg/kg (Q3W Regimen) (N=2) | PF-06647020 1.25 mg/kg (Q3W Regimen) (N=2) | PF-06647020 2.1 mg/kg (Q3W Regimen) (N=4) | PF-06647020 2.8 mg/kg (Q3W Regimen) (N=96) | PF-06647020 3.7 mg/kg (Q3W Regimen) (N=6) | PF-06647020 2.1 mg/kg (Q2W Regimen) (N=3) | PF-06647020 2.8 mg/kg (Q2W Regimen) (N=10) | PF-06647020 3.2 mg/kg (Q2W Regimen) (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06647020 0.2 mg/kg (Q3W Regimen) (N=2) | PF-06647020 0.5 mg/kg (Q3W Regimen) (N=2) | PF-06647020 1.25 mg/kg (Q3W Regimen) (N=2) | PF-06647020 2.1 mg/kg (Q3W Regimen) (N=4) | PF-06647020 2.8 mg/kg (Q3W Regimen) (N=96) | PF-06647020 3.7 mg/kg (Q3W Regimen) (N=6) | PF-06647020 2.1 mg/kg (Q2W Regimen) (N=3) | PF-06647020 2.8 mg/kg (Q2W Regimen) (N=10) | PF-06647020 3.2 mg/kg (Q2W Regimen) (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 17 | 2 | 0 | 2 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 30 | 2 | 0 | 4 | 4
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Macular oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 1 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 15 | 1 | 0 | 4 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 33 | 2 | 0 | 6 | 7
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 27 | 1 | 1 | 3 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 46 | 4 | 0 | 3 | 7
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 11 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 30 | 2 | 0 | 2 | 3
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 2 | 2 | 51 | 3 | 0 | 5 | 7
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 11 | 1 | 0 | 0 | 1
Breast cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 6 | 1 | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 9 | 1 | 0 | 2 | 3
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 7 | 2 | 0 | 4 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 30 | 2 | 1 | 5 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 21 | 0 | 0 | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 17 | 2 | 0 | 2 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 9 | 3 | 0 | 1 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 6 | 1 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 21 | 0 | 1 | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 7 | 1 | 0 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 9 | 0 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 17 | 1 | 1 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 3 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 6 | 1 | 0 | 1 | 4
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 35 | 3 | 0 | 4 | 7
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 1 | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 14 | 0 | 1 | 2 | 4
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 7 | 1 | 0 | 1 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 8 | 0 | 0 | 2 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 10 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 10 | 1 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 4 | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 41 | 3 | 3 | 8 | 7
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 9 | 1 | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 6 | 1 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 2
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid rash (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT02222922/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT02222922/SAP_001.pdf